CLINICAL TRIAL: NCT02947724
Title: The Use of Surgicel in Preventing Recurrence of Ovarian Endometriomas During Laparoscopic Surgery
Brief Title: Surgicel Reduces Ovarian Endometriomas Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 111949
Record Dates: First submitted 2016-10-21; First posted 2016-10-28 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Endometrioma
Keywords: chocolate cyst; laparoscopy; surgicel
MeSH Terms: conditions — Endometriosis | interventions — Surgicel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- drainage only (No Intervention): 50 patients underwent laparoscopic fenestration and electrocautery of the endometrioma cyst wall
- cystectomy only (No Intervention): 50 patients underwent laparoscopic excision of the endometrioma cyst wall
- drainage & Surgicel (Active Comparator): 50 patients underwent laparoscopic fenestration of the endometrioma cyst wall. Insertion of 4 pieces of SURGICEL® inside the cyst cavity
  Interventions: Drug: SURGICEL®
- cystectomy & Surgicel (Active Comparator): 50 patients underwent laparoscopic excision of the endometrioma cyst wall. Insertion of 4 pieces of SURGICEL® inside the remaining ovarian tissues.
  Interventions: Drug: SURGICEL®

INTERVENTIONS:
Drug: SURGICEL® — Insertion of 4 pieces of SURGICEL® inside the cyst cavity. Insertion of 4 pieces of SURGICEL® inside the remaining ovarian tissues.
  Arms: cystectomy & Surgicel; drainage & Surgicel

SUMMARY:
Two hundred women aged from 20 to 35 years undergoing conservative laparoscopic treatment of ovarian endometriomas (either by drainage or cyst wall excision) were included. Participants were randomized into 4 groups; group A (drainage only) in which 50 patients underwent laparoscopic fenestration and electrocautery of the endometrioma cyst wall, group B (cystectomy only) in which 50 patients underwent laparoscopic excision of the endometrioma cyst wall, group C (drainage & Surgicel) in which 50 patients underwent laparoscopic fenestration of the endometrioma cyst wall followed by insertion of 4 pieces of Surgicel inside the cyst cavity, group D (cystectomy & Surgicel) in which 50 patients underwent laparoscopic excision of the endometrioma cyst wall followed by insertion of 4 pieces of Surgicel inside the remaining ovarian tissues.All patients were followed up every 3 months for 2 years following the laparoscopic surgery. The primary outcome was the recurrence of endometriomas in the ipsilateral ovary (recurrence was defined as the presence of ovarian cysts with the characteristic sonographic features of endometriomas (≥1 cm). The ovarian reserve was reassessed (AMH & day 2 AFC) as a secondary outcome 6 months following the laparoscopy.

DETAILED DESCRIPTION:
Two hundred women aged from 20 to 35 years undergoing conservative laparoscopic treatment of ovarian endometriomas (either by drainage or cyst wall excision) were included. Participants were randomized into 4 groups; group A (drainage only) in which 50 patients underwent laparoscopic fenestration and electrocautery of the endometrioma cyst wall, group B (cystectomy only) in which 50 patients underwent laparoscopic excision of the endometrioma cyst wall, group C (drainage & Surgicel) in which 50 patients underwent laparoscopic fenestration of the endometrioma cyst wall followed by insertion of 4 pieces of Surgicel inside the cyst cavity, group D (cystectomy & Surgicel) in which 50 patients underwent laparoscopic excision of the endometrioma cyst wall followed by insertion of 4 pieces of Surgicel inside the remaining ovarian tissues. Randomization was done using computer generated random numbers.

Inclusion criteria included endometriosis-related clinical manifestations (infertility, pelvic pain or pelvic mass), unilateral & unilocular endometrioma (≥5 cm), rapidly growing endometrioma & good ovarian reserve (antimullerian hormone {AMH} > 1 ng/ml & antral follicular count {AFC} > 4). Recurrent & bilateral cases were excluded. In addition, patients who were unfit for surgery, suffered chronic diseases (e.g. cardiac disease or diabetes) or had any contraindication for laparoscopic surgery (excessive anterior abdominal wall scarring) were also excluded.

For all patients, full history was taken followed by complete physical examination & laboratory investigations (AMH & routine preoperative investigations). Day 2 transvaginal ultrasound (TVUS) was done using a 7.5 MHz vaginal probe of the General Electric Voluson E8 ultrasound unit (GE Healthcare Austria GmbH, Seoul, Korea) to confirm the presence and assess the size and side of the endometrioma (ovarian cyst with homogeneous low-level ground glass echogenicity of the cystic fluid) & to assess the AFC (Number of visible follicles from 2 to 10 mm) in both the affected and healthy ovary.

Cystectomy or drainage was done by one of the investigators. In cystectomy groups (B&D), a small window (2cm) was done in the cyst wall using diathermy followed by aspiration of the chocolate material from the cyst then stripping the cyst wall from ovarian tissue using 2 non-traumatic graspers (by traction-counter traction technique) and finally irrigating the remaining ovarian tissues with normal saline. In drainage groups (A & C), a small window (2cm) was done in the cyst wall using diathermy followed by aspiration of the chocolate material from the cyst & then irrigation of the cyst cavity with normal saline. In non-Surgicel groups (A&B), haemostasis & destruction of the remaining endometriotic cyst wall was done by bipolar electrocautery. In Surgicel groups (C&D), each SURGICEL® (oxidized regenerated cellulose - Ethicon US, LLC.) knitted fabric (5 x 10 cm) was divided into four equal pieces inserted inside the cavity of the cyst (group C) or the remaining ovarian tissues (group D). If the ovarian edges were gaped, approximation was done using 1-3 interrupted sutures of 4/0 polydioxanone (PDS® Suture - Ethicon US, LLC.). All patients were followed up every 3 months for 2 years following the laparoscopic surgery. The primary outcome was the recurrence of endometriomas in the ipsilateral ovary (recurrence was defined as the presence of ovarian cysts with the characteristic sonographic features of endometriomas (≥1 cm). The ovarian reserve was reassessed (AMH & day 2 AFC) as a secondary outcome 6 months following the laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis-related clinical manifestations (infertility, pelvic pain or pelvic mass)
* Unilateral & unilocular endometrioma (≥5 cm),
* Rapidly growing endometrioma
* Good ovarian reserve (antimullerian hormone {AMH} > 1 ng/ml & antral follicular count {AFC} > 4).

Exclusion Criteria:

* Recurrent & bilateral cases
* Patients who were unfit for surgery, suffered chronic diseases (e.g. cardiac disease or diabetes)
* PATIENTS had any contraindication for laparoscopic surgery (excessive anterior abdominal wall scarring) .

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
recurrence of endometriomas in the ipsilateral ovary | 2 YEARS
  recurrence was defined as the presence of ovarian cysts with the characteristic sonographic features of endometriomas (≥1 cm)

SECONDARY OUTCOMES:
biochemical ovarian reserve | 6 months after laparoscopy
  serum antimullerian hormone measuremnt
ultrasonographic ovarian reserve | 6 months following the operation
  antral follicle count on day 2 using transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: moutaz elsherbini, MD, Principal Investigator — Assistant professor of obstetrics and gynecology - Cairo university
Locations (1):
- Kasr Elainy Hospital (Cairo University), Cairo, Egypt

REFERENCES:
- [Derived] Shaltout MF, Elsheikhah A, Maged AM, Elsherbini MM, Zaki SS, Dahab S, Elkomy RO. A randomized controlled trial of a new technique for laparoscopic management of ovarian endometriosis preventing recurrence and keeping ovarian reserve. J Ovarian Res. 2019 Jul 20;12(1):66. doi: 10.1186/s13048-019-0542-0. PMID 31325962